CLINICAL TRIAL: NCT04274153
Title: A Pilot Study of the Immunogenicity of a Two-dose Protocol for 9-valent Human Papilloma Virus Vaccination in Postpartum Girls and Women (15-45 Years Old) Previously Unvaccinated Against HPV
Brief Title: HPV Vaccination Study in Postpartum Women
Acronym: PPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00227941
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: HPV; Immunization; Human Papilloma Virus
Keywords: Human Papilloma Virus; HPV; Immunization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gardasil9 (Experimental): Two doses of the 9-valent HPV vaccine to be administered to participants at 0 and 6 months. Additional HPV vaccine dose will be offered after final blood draw at 12 months.
  Interventions: Biological: Gardasil9

INTERVENTIONS:
Biological: Gardasil9 — Two doses of the HPV vaccine across a 12 month period (two doses of 0.5mL).

SUMMARY:
The human papillomavirus (HPV) is the most common sexually transmitted infection (STI) in the United States (U.S.) and is responsible for a wide range of conditions, including cancers within the anogenital tract and the oropharynx. In just the U.S. alone, it's estimated that HPV causes 330,000 cases of precancerous cervical dysplasia and 12,000 cases of cervical cancer. The investigators propose a 2-dose HPV vaccination study in women seeking postpartum care at Johns Hopkins University. The investigators will measure the immunogenicity and acceptability of the vaccine in the postpartum setting.

DETAILED DESCRIPTION:
This is a pilot, non-inferiority clinical trial using historical controls. Participants will have whole blood drawn at 0 months, 6 months, and 7 months and receive the HPV vaccine at 0 months, 6 months, and 12 months. Each blood draw will consist of one 15mL red top tube to measure HPV serologies and hormone levels. All blood samples collected will be analyzed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants biologically born as females between the ages of 15 through 45 who have delivered a live born baby within the past 72 hours.

Exclusion Criteria:

* Pregnancy
* Severe allergic reaction to vaccine components
* Prior receipt of an HPV vaccine dose
* Fetal demise or stillbirth
* Allergy to latex or yeast
* Moderate or severe acute illness (deemed by the investigator to exclude)
* Immunosuppression (e.g., HIV, solid organ transplant).

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women seeking postpartum care at Johns Hopkins University who self-report never receiving an HPV vaccination.
Enrollment: 225 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenell Coleman, MD, Principal Investigator — Johns Hopkins University; Chailee Moss, MD, Principal Investigator — Johns Hopkins University; Betty Chou, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Derived] Moss CF, Wang R, Sao S, Chou B, Perin J, Lander ME, Thaker SM, Mann M, Coleman JS. Immunogenicity of 2-Dose HPV Vaccine Series for Postpartum Women: An Open-Label, Nonrandomized, Noninferiority Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352996. doi: 10.1001/jamanetworkopen.2023.52996. PMID 38285445

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gardasil9
Started | 225
Completed | 169
Not Completed | 56

BASELINE CHARACTERISTICS:
Arm/Group | Gardasil9
Number analyzed (Participants) | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic/Latino | 134
  Race/Ethnicity: Black/African American | 43
  Race/Ethnicity: Asian | 9
  Race/Ethnicity: White/Caucasian | 36
  Race/Ethnicity: Two or more races | 2
  Race/Ethnicity: Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 225
Highest level of education [Count of Participants; unit: Participants]
  Grade 11 or less | 71
  Grade 12 to some college | 99
  Bachelor's degree or higher | 55
Employed [Count of Participants; unit: Participants]
  Yes | 74
  No | 151

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of a Two-dose 9-valent HPV Vaccination as Assessed by Antibody Titer
Description: Measure the immunogenicity of a two-dose 9-valent HPV vaccination regimen in postpartum women previously unvaccinated against the HPV 16 virus. Immunogenicity will be assessed by the antibody responses. The Geometric mean titers will be measured using milli Merck units (mMU)/mL.
Time Frame: Up to 23 months
Population: We excluded participants whose anti-HPV 16 titer was above the seroconversion limit and the baseline. Therefore, only 129 were included in this analysis
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Gardasil9
Number analyzed (Participants) | 129
mMU/mL | 7177.6 [6041.0 to 8528.0]

2. Secondary Outcome: Antibody Response to the Other 8 HPV Types
Description: The antibody types that will be measured are HPV types 6, 11, 18, 31, 33, 45, 52, and 58.
  The milli Merck units (mMU)/mL of measure will be used to determine antibody response.
Time Frame: Up to 23 months
Population: During analysis, we exclude participants who had antibodies titers above the seroconversion limit at the baseline for each HPV subtype seperately. Therefore, the number of participants analyzed are smaller than 225.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Gardasil9
Number analyzed (Participants) | 133
mMU/mL
  6 | 2187.2 [1861.3 to 2570.2]
  11 | 1492.1 [1289.1 to 1727.1]
  18 | 1589.8 [1333.6 to 1895.2]
  31 | 1077.5 [924.8 to 1255.4]
  33 | 792.8 [680.0 to 924.4]
  45 | 323.2 [278.9 to 374.6]
  52 | 582.9 [512.2 to 663.3]
  58 | 802.8 [681.9 to 945.1]

3. Secondary Outcome: Seropositivity for HPV 16 After 1-dose
Description: Calculate the percentage of participants that seroconverted.
Time Frame: After the first dose, up to 7 months
Population: There were some participants seroconverted at the baseline so were excluded from the analysis for each type of HPV.
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 134
Participants | 118

4. Secondary Outcome: Seropositivity for HPV 16 After 2-doses
Description: Calculate the percentage of participants that seroconverted.
Time Frame: After the second dose, up to 2 months
Population: Participants with anti-HPV 16 titer above the seropositivity threshold were excluded in this analysis. This is analysis among participants who received the second dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 128
Participants | 128

5. Secondary Outcome: Percentage of Participants With Baseline Titers Suggestive of Natural Inoculation or Prior Vaccination to HPV 16
Description: Running an assay to measure a participants natural inoculation or prior vaccination before administration of the 1st dose.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 225
Participants | 91

6. Secondary Outcome: Percentage of Participants Who Complete 2-dose Vaccination
Description: Calculate the amount of participants that complete 2-dose vaccination.
Time Frame: At the end of the study, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 225
Participants | 174

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Gardasil9
All-Cause Mortality (participants affected / at risk) | 0/225
Serious Adverse Events (participants affected / at risk) | 0/225
Other Adverse Events (participants affected / at risk) | 1/225
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gardasil9 (N=225)
Not serious adverse event due to medication (Skin and subcutaneous tissue disorders) | 1 — Participant's arm was swollen and painful for several days after receiving her second dose of the HPV vaccine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT04274153/Prot_SAP_000.pdf